CLINICAL TRIAL: NCT00431145
Title: Influence of Combined Therapy of Niacin and Statins on Stem Cell Mobilization and Inflammatory Parameters in Patients Suffering From Coronary Artery Disease - Randomized Clinical Study -
Brief Title: Niacin As Secondary Prevention Of Coronary Artery Disease (NASPOCAD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20091977
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2007-02-05 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Niacin

INTERVENTIONS:
Drug: Niacin
Drug: Niacin+Statin

SUMMARY:
Aim of the study is to show additional effects of the combined therapy of niacin and statins analyzing number and function of EPCs and other stem cell populations and adiponectin as well as hsCRP levels in patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old, male or female
* Have stable coronary artery disease (i.e. no acute event like myocardial infarction or PTCA less then 3 months ago)
* LDL > 100 mg/dl
* HDL < 50 mg/dl
* Triglycerides < 400 mg/dl
* No Nicotine abuse for at least 3 months
* Statin-therapy for more than 4 weeks
* Give a written informed consent
* Have the ability to understand the requirements of the study, and agree and be able to return for the required assessments.

Exclusion Criteria:

* Women of childbearing potential, pregnancy or being lactating
* Current participation in another clinical trial
* Have other severe concurrent illness (e.g., active infection, malignancy)
* Have a history of alcohol or drug abuse within 3 months of admission or factors making follow-up difficult or unlikely.
* Have significant or unexplained liver dysfunction or chronic increased levels of transaminases (ALT, AST)
* Suffer from myopathy, active peptic disease or arterial bleeding
* Have a known hypersensitivity against niacin or statins
* Are actually treated with any of itraconazole, ketoconazole, HIV-Protease-Inhibitors, erythromycin, clarithromycin, telithromycin, nefazodone.
* Actual therapy with ezetimibe
* Diabetes mellitus Type I

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-10

PRIMARY OUTCOMES:
numbers of EPCs and inflammatory markers
adiponectin
hsCRP
each after 8 weeks

SECONDARY OUTCOMES:
numbers of EPCs,
inflammatory markers
adiponectin
hsCRP
each after 4 weeks
number and type of progenitor cells
dendritic cells
cytokines
lipoproteins in peripheral blood
vascular function
each after 4 and 8 weeks
carotid artery distensibility
carotid artery plaque composition
each after 8 weeks
optionally 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang M Franz, MD, Principal Investigator — University of Munich/Germany
Locations (1):
- University of Munich, Munich, Germany